CLINICAL TRIAL: NCT02189226
Title: Usefulness of Probe-based Confocal Laser Endo-microscopy in Delineation of Margin of Early Gastric Cancer for Endoscopic Submucosal Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2013-0009
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Last update posted 2019-04-01 (Actual); Status verified 2015-12

CONDITIONS: Early Gastric Cancer
Keywords: probe-based confocal laser endomicroscopy (pCLE), early gastric cancer (EGC), endoscopic submucosal dissection (ESD), margin
MeSH Terms: conditions — Stomach Neoplasms; Margins of Excision | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- probe-based confocal laser endomicroscopy (pCLE) group (Experimental)
  Interventions: Device: Endoscopic submucosal dissection (ESD) with or without probe-based confocal laser endomicroscopy (pCLE)
- chromoendoscopy (CE) group (Active Comparator)
  Interventions: Device: Endoscopic submucosal dissection (ESD) with or without probe-based confocal laser endomicroscopy (pCLE)

INTERVENTIONS:
Device: Endoscopic submucosal dissection (ESD) with or without probe-based confocal laser endomicroscopy (pCLE) — Before ESD, the lesion will be observed either by pCLE or by CE to determine proximal and distal margin of the lesion. In the pCLE group, after injection of intravenous fluorescein, the lesion will be observed using a flexible confocal miniprobe. In the CE group, the lesion will be observed conventionally under white light after spraying indigocarmine directly via the forceps channel. Marking dots will be placed on both margins using needle knife. Then several dots will be marked on the surrounding normal mucosa 5 mm from the tumor with Argon plasma coagulation. After injection of saline solution with epinephrine into the submucosa, an initial cut will be made with needle knife outside the line of surrounding marks. An insulation-tipped (IT) knife will be inserted into initial cut, and electrosurgical current will be applied to complete the incision around the tumor. After the circumferential cut, the submucosa will be dissected with the IT knife.

SUMMARY:
The aim of this study is to evaluate the usefulness of pCLE (probe-based confocal laser endomicroscopy) compared with conventional chromoendoscopy (CE) for delineating the margin of early gastric cancer (EGC) with endoscopic submucosal dissection (ESD).

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients diagnosed as EGC and treated by ESD with following criteria:1) Differentiated mucosal cancer without ulcer 2) Differentiated mucosal cancer with ulcer, ≤ 3 cm 3) Differentiated minute (<500 μm) submucosal invasive cancer, ≤ 3 cm 4) Undifferentiated mucosal cancer without ulcer, ≤ 2 cm
* Consecutive patients diagnosed as low- and high-grade dysplasia with suspicion of EGC and treated by ESD

Exclusion Criteria:

* Coagulopathy : International normalized ratio [INR] > 1.5 or platelet count <50,000 cell/cubic millimeter)
* Impaired renal function : Cr > 1.2 mg/dL
* Pregnancy or breast-feeding
* Age < 20 years
* Allergy to fluorescein dye
* Inability to provide informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01-20 (Actual); Study Completion 2015-01-20 (Actual)

PRIMARY OUTCOMES:
Complete resection rate | One week after ESD
  Complete resection is defined as en bloc resection with negative horizontal, vertical margin and distance from marking dot to histologic margin will be measured.

SECONDARY OUTCOMES:
Horizontal cut end-positive | Within the first 30 days after ESD
vertical cut end-positive | Within the first 30 days after ESD
procedure time | 1 day
adverse event | Within the first 30 days after ESD

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea